CLINICAL TRIAL: NCT01619852
Title: The Effect of Lidocaine to Prevent the Development of Chronic Post-Surgical Pain
Brief Title: Lidocaine and Prevention of Chronic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Gildasio De Oliveira, Principal Investigator, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: STU00061676
Record Dates: First submitted 2012-06-12; First posted 2012-06-14 (Estimated); Results first posted 2019-11-27 (Actual); Last update posted 2019-11-27 (Actual); Status verified 2019-11

CONDITIONS: Surgery
Keywords: Surgery; Breast; Pain; Chronic Pain; Lidocaine; Anesthesia; Gynecologic; Urologic
MeSH Terms: conditions — Pain; Chronic Pain | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group L (Active Comparator): Group L will receive a 1.5 mg/kg bolus of intravenous lidocaine followed by a 2mg/kg/hr infusion that will be started at the time of surgical induction and will be discontinued one hour after the end of the surgical procedure.
  Interventions: Drug: Group L (lidocaine)
- .9% normal saline placebo (Placebo Comparator): .9% normal saline administered as a bolus then as a maintenance infusion for the length of the surgical case.
  Interventions: Drug: .9 normal saline placebo

INTERVENTIONS:
Drug: .9 normal saline placebo — Administration of .9 normal saline placebo as a bolus and as maintenance throughout the length of the surgical procedure.
  Arms: .9% normal saline placebo
Drug: Group L (lidocaine) — Group L will receive a 1.5 mg/kg bolus of intravenous lidocaine followed by a 2mg/kg/hr infusion that will be started at the time of surgical induction and will be discontinued one hour after the end of the surgical procedure.
  Arms: Group L

SUMMARY:
The study seeks to investigate a safe and inexpensive strategy to reduce persistent post-surgical pain that can affect up to 60% of patients undergoing surgical procedures.

Hypotheses: Perioperative systemic lidocaine reduces the persistence of chronic pain in patients undergoing surgical procedures.

DETAILED DESCRIPTION:
After approval from Northwestern University's IRB, female subjects undergoing urologic, gynecologic or breast surgery will be included in the study. Informed consent will be obtained from all participants. Subject will be randomized using a computer generated table of random numbers into two groups: Group L will receive a 1.5 mg/kg bolus of intravenous lidocaine followed by a 2mg/kg/hr infusion that will be started at the time of surgical induction and will be discontinued one hour after the end of the surgical procedure. Group P will receive the same amount of saline in the same fashion. This dose regimen of systemic lidocaine chosen in the current study has been consistently associated with a reduction of acute postoperative pain.4 There will be no visual characteristic differences between any of the infusions studied and they will all be labeled as a study drug. Patients will receive a standard anesthetic regimen consisting of propofol, fentanyl, succinylcholine, and sevoflurane. Patients will receive ondansetron 4mg and dexamethasone 4 mg to prevent postoperative nausea and vomiting. They will also receive 10 mcg/kg of hydromorphone at the end of surgery to prevent postoperative pain. In the PACU, patients will receive additional doses of hydromorphone to keep pain <4/10 (on a scale where 0 means no pain and 10 is the worst pain possible). On PACU discharge, patients will receive a patient-controlled IV hydromorphone analgesia pump set at 0.2mg IV bolus, no basal infusion and a lockout time of 15 minutes. The intraoperative and postoperative data (pain scores, opioid consumption, side effects) will be collected by a research assistant blinded to the group allocation). Other data collection variables include : Preoperative (Age, BMI, ethnicity, comorbidities, preoperative medication(s), psychiatric disease, pain in the operative area, pain at other locations), Intraoperative (description of surgical procedure, surgical duration, surgical procedure on nerve areas, preservation of the nerves in the operative area nerve, indication for the surgical procedure, intraoperative opioids dose, and Postoperative pain instruments (evaluation of early pain, twenty four hour opioid consumption, drugs and other treatments used in the postoperative period.

QOR 40 questionnaire will be completed by the participant at 24 hours after surgery if they have not been discharged from the hospital. If they have been discharged, the research assistant will contact the participant by telephone to complete the questionnaire.

Patients will be evaluated for the presence and severity of chronic pain as well as the quality of life impact of pain at baseline, three and six months after surgery using a validated instrument in accordance with the IMMPACT recommendations to assess chronic pain and its impact on the patient's quality of life (Brief pain Inventory).8 To characterize the chronic pain, both the short form McGill pain questionnaire and the Modified LANNS scale will be also administered at three and six months.9,10 If there is no response to the 3 month questionnaire, the subject will be contacted by telephone to complete the questionnaire.

Subjects who are experiencing suicidal ideation will be referred to Northwestern Memorial Hospital Emergency Department. The primary care surgeon will also be notified by the principal investigator. Mood will be assessed using the Beck Depression Inventory.14

ELIGIBILITY:
Inclusion Criteria:

* Age 18-64,
* Females undergoing gynecological, urological or breast surgery

Exclusion Criteria:

* pregnant,
* history of chronic use of opioids,
* allergy to local anesthetics,
* history of cardiac arrhythmias Drop out: patient or surgeon request

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 148 (Actual)
Dates: Start 2012-06; Primary Completion 2014-07 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gildasio De Oliveira, M.D., Principal Investigator — Northwestern University
Locations (1):
- Prentice Womens' Hospital, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] 1) Eric J. Visser. Chronic post-surgical pain: Epidemiology and clinical implications for acute pain management. Acute Pain.2006:8; 73-81
- [Background] Phillips CJ, Harper C. The economics associated with persistent pain. Curr Opin Support Palliat Care. 2011 Jun;5(2):127-30. doi: 10.1097/SPC.0b013e3283458fa9. PMID 21430542
- [Background] Amr YM, Yousef AA. Evaluation of efficacy of the perioperative administration of Venlafaxine or gabapentin on acute and chronic postmastectomy pain. Clin J Pain. 2010 Jun;26(5):381-5. doi: 10.1097/AJP.0b013e3181cb406e. PMID 20473044
- [Background] Vigneault L, Turgeon AF, Cote D, Lauzier F, Zarychanski R, Moore L, McIntyre LA, Nicole PC, Fergusson DA. Perioperative intravenous lidocaine infusion for postoperative pain control: a meta-analysis of randomized controlled trials. Can J Anaesth. 2011 Jan;58(1):22-37. doi: 10.1007/s12630-010-9407-0. PMID 21061107
- [Background] Attal N, Gaude V, Brasseur L, Dupuy M, Guirimand F, Parker F, Bouhassira D. Intravenous lidocaine in central pain: a double-blind, placebo-controlled, psychophysical study. Neurology. 2000 Feb 8;54(3):564-74. doi: 10.1212/wnl.54.3.564. PMID 10680784

RESULTS

PARTICIPANT FLOW:
Groups:
- Lidocaine (Group L): Lidocaine (Group L) will receive a 1.5 mg/kg bolus of intravenous lidocaine followed by a 2mg/kg/hr infusion that will be started at the time of surgical induction and will be discontinued one hour after the end of the surgical procedure.
Period: 24 Hour Assessment
Arm/Group | Lidocaine (Group L) | .9% Normal Saline Placebo
Started | 75 | 75
Completed | 74 | 74
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1
Period: 3 Month Follow up
Arm/Group | Lidocaine (Group L) | .9% Normal Saline Placebo
Started | 74 | 74
Completed | 43 | 40
Not Completed | 31 | 34
Not completed — Lost to Follow-up | 31 | 34

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group L | .9% Normal Saline Placebo | Total
Number analyzed (Participants) | 75 | 75 | 150
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 75 | 75 | 150
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75 | 75 | 150
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  White | 58 | 60 | 118
  African American | 12 | 10 | 22
  Asian | 2 | 3 | 5
  Hispanic | 2 | 2 | 4
  Other | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 75 | 75 | 150
Body Mass Index (BMI) [Mean (Full Range); unit: kg/mg^2] — BMI =(weight in kilograms) / height in meters²
  kg/mg^2 | 24 [21 to 29] | 25 [22 to 30] | 24.5 [21 to 30]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Chronic Persistent Pain 3 Months After Surgery as Determined by Character Severity (Yes/no).
Description: The participants development of chronic persistent pain 3 months after surgery as determined by character severity (yes/no).
Time Frame: 3 months
Measure: Number; unit: participants
Arm/Group | Group L | .9% Normal Saline Placebo
Number analyzed (Participants) | 43 | 40
participants | 2 | 6
Statistical Analysis 1: Comparison: Group L vs .9% Normal Saline Placebo; Test type: Superiority or Other; p = .19, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Quality of Recovery
Description: Quality of recovery (QoR-40 instrument) is a 40-item questionnaire that provides a global score and sub-scores across five dimensions: patient support, comfort, emotions, physical independence, and pain. Score range: 40 to 200. A score of 40 demonstrates poor recovery and a maximum score of 200 represents good recovery. The higher the score the better recovery after surgery.
Time Frame: 24 hours post operative
Measure: Median (Inter-Quartile Range); unit: units on a scale
Groups:
- Lidocaine (Group L): Lidocaine (Group L) will receive a 1.5 mg/kg bolus of intravenous lidocaine followed by a 2mg/kg/hr infusion that will be started at the time of surgical induction and will be discontinued one hour after the end of the surgical procedure.
  Lidocaine (Group L): will receive a 1.5 mg/kg bolus of intravenous lidocaine followed by a 2mg/kg/hr infusion that will be started at the time of surgical induction and will be discontinued one hour after the end of the surgical procedure.
Arm/Group | Lidocaine (Group L) | .9% Normal Saline Placebo
Number analyzed (Participants) | 74 | 74
units on a scale | 158 [147 to 178] | 169 [151 to 176]
Statistical Analysis 1: Comparison: Lidocaine (Group L) vs .9% Normal Saline Placebo; Test type: Superiority or Other; p = 0.64, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Post-surgical Persistent Pain Using Validated Questionnaires (S-LANNS Questionnaire, McGill Questionnaire, Brief Pain Inventory) to Assess Pain Qualities in Accordance With IMMPACT Recommendations.
Description: The development of chronic pain 3 months after surgery determined by the Leads Assessment of Neuropathic Symptoms and Signs (LANSS) scale, a valid 7-item tool for identifying patients whose pain is dominated by neuropathic mechanisms. Each item is a binary response (yes or no) to the presence of symptoms (5 items) or clinical signs (2 items), range 0-24 points. A score ≥ 12, neuropathic mechanisms are likely to be contributing to the patient's pain. A score < 12 is unlikely to be contributing. McGill questionnaire (Sensory domain) - 11 descriptors rated on an intensity scale as 0=none, 1=mild, 2=moderate, 3=severe. The higher the score, greater the pain (range 0-33). McGill questionnaire (Motivational-affective) 4 affect descriptors rated on an intensity scale as 0=none, 1=mild, 2=moderate, 3=severe.The higher the score the greater the pain (range 0-12) Brief pain inventory - pain severity (0, no pain, 10 excruciating pain); Greater the score; greater the pain (range 0-10).
Time Frame: 3 months
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Group L | .9% Normal Saline Placebo
Number analyzed (Participants) | 43 | 40
units on a scale
  S-LANNS | 3 [0 to 10] | 3 [0 to 8]
  McGill Questionaire-Sensory Discrimation | 4 [1 to 7] | 3 [1 to 7]
  McGill Questionaire-Motivational-affective | 0 [0 to 1] | 0 [0 to 2]
  Brief Pain Inventory | 1 [0 to 3] | 1 [0 to 3]
Statistical Analysis 1: Comparison: Group L vs .9% Normal Saline Placebo; Test type: Superiority or Other; p = 0.68, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Group L vs .9% Normal Saline Placebo; McGill Questionnaire-Sensory-discriminative dimension; Test type: Superiority or Other; p = 0.69, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Group L vs .9% Normal Saline Placebo; McGill Questionnaire-affective dimension; Test type: Superiority or Other; p = 0.75, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Group L vs .9% Normal Saline Placebo; Brief Pain Inventory; Test type: Superiority or Other; p = 0.81, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Opioid Consumption
Description: The amount of opioid analgesics consumed was converted to an equivalent dose of intravenous morphine.
Time Frame: 24 hours
Measure: Median (Inter-Quartile Range); unit: equivalent dose of intravenous morphine
Arm/Group | Group L | .9% Normal Saline Placebo
Number analyzed (Participants) | 74 | 74
equivalent dose of intravenous morphine | 34 [17 to 46] | 39 [21 to 57]
Statistical Analysis 1: Comparison: Group L vs .9% Normal Saline Placebo; Test type: Superiority or Other; p = .19, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Postoperative Pain
Description: Postoperative pain within the first 24 hours. Area under the numeric rating scale for pain versus time curve during the first 24 hours after surgery (score * hr). Numeric rating scale for pain on a scale of 0-10 (0 is no pain and 10 is high pain) versus time curve during the first 24 hours ( score * hr). The pain scores were collected upon arrival to recovery area, 30 minutes, 1 hour and every 6 hours up to 24 hours following the procedure. Minimum score is 60, Maximum score is 170. A higher value indicates more pain.
Time Frame: 24 hours
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Group L | .9% Normal Saline Placebo
Number analyzed (Participants) | 74 | 74
score on a scale | 116 [88 to 142] | 119 [91 to 148]
Statistical Analysis 1: Comparison: Group L vs .9% Normal Saline Placebo; Test type: Superiority or Other; p = .29, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 24 hours after surgery completion.
Arm/Group | Group L | .9% Normal Saline Placebo
Serious Adverse Events (participants affected / at risk) | 0/74 | 0/74
Other Adverse Events (participants affected / at risk) | 0/74 | 0/74

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No